CLINICAL TRIAL: NCT01865851
Title: Comparison of the Classic Face Mask Versus NuMask for Preoxygenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nimmagadda, Usharani, M.D. (Individual)
Responsible Party: Principal Investigator, Usharani Nimmagadda, Anesthesiologist, Advocate Illinois Masonic Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB5558
Record Dates: First submitted 2013-05-14; First posted 2013-05-31 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Inspired Oxygen (FIO2), End-tidal Oxygen (ETO2), End-tidal Carbon Dioxide (ETCO2) and Respiratory Rate (RR) Will be Measured Every 30 Seconds
Keywords: Inspired oxygen; end-tidal oxygen; end-tidal carbon dioxide; respiratory rate; preoxygenation; classic face mask; NuMask

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Start with Classic Face Mask Group (Active Comparator): The volunteers will be asked to breathe normally (Tidal Volume Breathing) through face mask for 5 minutes. After 5 minutes, the volunteers will be asked to breathe room air for 5 minutes and then breathe through a NuMask for 5 minutes. This will be followed by room air breathing for 5 minutes. At the end of the 5 minutes of room air breathing, the same volunteers will be asked to breathe through the face mask for 5 minutes.
  Interventions: Device: Classic Face Mask and NuMask
- Start with NuMask Group (Active Comparator): The volunteers will be asked to breathe through the NuMask for 5 minutes, followed by room air breathing for 5 minutes, then 5 minutes of breathing through the face mask. This will be followed by room air breathing for 5 minutes and then 5 minutes of NuMask breathing.
  Interventions: Device: Classic Face Mask and NuMask

INTERVENTIONS:
Device: Classic Face Mask and NuMask

SUMMARY:
Currently used face mask has certain disadvantages; such as, not providing a complete seal in certain patients, causing hand fatigue after holding the mask in place for more than a few minutes, causing claustrophobia in an occasional patient, the need to hold the mask from head of the bed, and possible worsening of the trauma in patients with facial injuries, and the need to use different size masks in different patients. The NuMask overcomes all of these disadvantages and does benefit the patients.

DETAILED DESCRIPTION:
The administration of oxygen before anesthetic induction and tracheal intubation (preoxygenation) is a well-recognized technique designed to increase oxygen reserves and thereby delay the onset of arterial oxygen desaturation during apnea. It is particularly important if manual ventilation is not desirable prior to intubation (eg: rapid sequence induction) or if difficulty with ventilation or intubation is anticipated or in patients with oxygen transport limitations. Because the "cannot ventilate/cannot intubate" situation is an unpredictable event, theoretically all patients should be maximally preoxygenated.

Fraction of inspired oxygen (FIO2) is one of the factors in achieving maximal preoxygenation. A common reason for the failure to achieve an FIO2 close to 1.0 is a leak under the face mask. Several factors may contribute to the leak. These are edentulous patients, patients with sunken cheeks, bearded patients, the presence of nasogastric tubes, wrong size face masks, improper use of head straps, and patients with large heads and faces where even the large size mask may not fit properly.

Recently a new intraoral mask "NuMask" has become available for anesthetic induction. It is placed under the lips and outside the gums of the patient mouth (similar to snorkel mouth piece), thus providing a good seal in almost any patient. In addition to providing a good seal, the NuMask has other advantages over the standard face mask. It has very small dead space (18 cc : 110 cc), provides comfortable grip, ventilation can be provided from any position and causes less facial trauma.

The efficacy of preoxygenation using the NuMask will be compared to the classic face mask in approximately 30 healthy and consenting adult volunteers. All of the volunteers will be randomly assigned into one of 2 groups. All volunteers will be tested for three (3) periods of 5 minute intervals. Inspired oxygen (FIO2), end-tidal oxygen (ETO2), end-tidal carbon dioxide (ETCO2) and respiratory rate (RR) will be tested. Analysis of the data may reveal whether the NuMask is equal, superior, or inferior to the classic face mask in achieving maximal preoxygenation.

Although the NuMask has been tested and used in various scenarios of airway management, its efficacy in achieving maximal preoxygenation has not been studied

ELIGIBILITY:
Inclusion Criteria:

* volunteers

Exclusion Criteria:

* under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Inspired (FIO2) | 30 minutes
  Healthy volunteers will be randomly breathing 100% oxygen through either a classic face mask or NuMask for 5 minutes. Measurements will be taken every 30 seconds. The purpose of the study is to evaluate which mask will provide maximal pre-oxygenation (more than 90% end-tidal oxygen).

SECONDARY OUTCOMES:
ETCO2 | 30 minutes
ETO2 | 30 minutres
Respiratory Rate | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nick Knezevic, PhD, MD, Study Director — Advocate Illinois Masonic Medical Center, Department of Anesthesiology
Locations (1):
- Advocate Illinois Masonic Medical Center, Department of Anesthesia, Chicago, Illinois, United States

REFERENCES:
- [Result] Nimmagadda U, Salem MR, Joseph NJ, Miko I. Efficacy of preoxygenation using tidal volume and deep breathing techniques with and without prior maximal exhalation. Can J Anaesth. 2007 Jun;54(6):448-52. doi: 10.1007/BF03022030. PMID 17541073
- [Result] Nimmagadda U, Chiravuri SD, Salem MR, Joseph NJ, Wafai Y, Crystal GJ, El-Orbany MI. Preoxygenation with tidal volume and deep breathing techniques: the impact of duration of breathing and fresh gas flow. Anesth Analg. 2001 May;92(5):1337-41. doi: 10.1097/00000539-200105000-00049. PMID 11323373
- [Result] Nimmagadda U, Salem MR, Joseph NJ, Lopez G, Megally M, Lang DJ, Wafai Y. Efficacy of preoxygenation with tidal volume breathing. Comparison of breathing systems. Anesthesiology. 2000 Sep;93(3):693-8. doi: 10.1097/00000542-200009000-00018. PMID 10969302
- [Result] Ramez Salem M, Joseph NJ, Crystal GJ, Nimmagadda U, Benumof JL, Baraka A. Preoxygenation: comparison of maximal breathing and tidal volume techniques. Anesthesiology. 2000 Jun;92(6):1845-7. No abstract available. PMID 10839945